CLINICAL TRIAL: NCT03383692
Title: A Phase 1, Multicenter, Open-label, Single Sequence Crossover Study to Evaluate Drug-drug Interaction Potential of OATP1B/CYP3A Inhibitor on the Pharmacokinetics of DS-8201a in Subjects With HER2-expressing Advanced Solid Malignant Tumors
Brief Title: Study of DS-8201a for Participants With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-A104; 173790 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2017-12-07; First posted 2017-12-26 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-09

CONDITIONS: Neoplasm Metastasis
Keywords: Unresectable or metastatic solid malignant tumors; Solid malignant tumors; Oncology; HER2; Antibody drug conjugate; ADC
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — trastuzumab deruxtecan; Ritonavir; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: DS-8201a + Ritonavir (Experimental): DS-8201a will be administered as an intravenous (IV) solution once every 3 weeks (Q3W) + Ritonavir twice daily (BID) on Day 17 of Cycle 2 until Day 21 of Cycle 3
  Interventions: Drug: DS-8201a; Drug: Ritonavir
- Cohort 2: DS-8201a + Itraconazole (Experimental): DS-8201a will be administered as an intravenous (IV) solution once every 3 weeks (Q3W) + Itraconazole BID on Day 17 of Cycle 2 followed by 200 mg daily (QD) until Day 21 of Cycle 3
  Interventions: Drug: DS-8201a; Drug: Itraconazole

INTERVENTIONS:
Drug: DS-8201a — DS-8201a is provided as a sterile lyophilized powder of DS-8201a in a glass vial, which will be dissolved and administered as an intravenous (IV) solution
Drug: Ritonavir — Ritonavir is a OATP1B inhibitor; an antiretroviral tablet for oral administration
  Other Names: Norvir
  Arms: Cohort 1: DS-8201a + Ritonavir
Drug: Itraconazole — Itraconazole is a CYP3A inhibitor; an antifungal tablet for oral administration
  Other Names: Sporanox; Orungal
  Arms: Cohort 2: DS-8201a + Itraconazole

SUMMARY:
HER2-positive cancer is a cancer that tests positive for a protein called human epidermal growth factor receptor 2 (HER2). HER2 promotes the growth of certain cancer cells. This study will test an experimental drug called DS-8201a that has not been approved by the health authorities yet.

DS-8201a will be tested for safety in patients with advanced solid malignant tumors that test positive for HER2. It also will test how DS-8201a moves within the body (pharmacokinetics).

DETAILED DESCRIPTION:
The expected time from the first subject's enrollment until the last subject's enrollment is approximately 8.5 months. The screening period is 28 days and each cycle of treatment is 21 days.

The data for the primary analysis will cutoff after all subjects have either discontinued the study or completed at least 3 cycles, whichever comes first. After the primary analysis, the main study will be closed and transition to the extension period.

Depending on the preliminary results of Cohort 1, Sponsor may decide whether Cohort 2 will be opened or not.

The number of treatment cycles is not fixed in this study. Subjects who continue to derive clinical benefit from the study drug in the absence of withdrawal of consent, progressive disease (PD), or unacceptable toxicity may continue the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically documented unresectable or metastatic solid malignant tumor, with HER2 expression [immunohistochemistry (IHC) 3+, 2+, or 1+ and/or in situ hybridization (ISH) +], Next Generation Sequencing, or other analysis techniques as appropriate] that is refractory to or intolerable with at least one prior systemic chemotherapy regimen, or for which no standard treatment is available
* Has a left ventricular ejection fraction (LVEF) ≥ 50%
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1

Exclusion Criteria:

* Has a contraindication for receiving ritonavir or itraconazole according to the prescribing information
* Has a medical history of myocardial infarction within 6 months before enrollment or symptomatic congestive heart failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (10):
- Japan (7):
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Nagaizumicho, Shizuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Takahashi S, Bando H, Kinoshita I, Modi S, Tsurutani J, Bang YJ, Sato Y, Nakatani S, Lee C, Sugihara M, Okuda Y, Iwata H. Trastuzumab deruxtecan in patients with human epidermal growth factor receptor 2-expressing salivary gland carcinoma: a pooled analysis of two phase I studies. Jpn J Clin Oncol. 2024 Apr 6;54(4):434-443. doi: 10.1093/jjco/hyad181. PMID 38231777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants who met all inclusion criteria and no exclusion criteria were enrolled and received treatment at 10 study centers in Japan, South Korea, and Taiwan.
Pre-assignment Details: Based on the pharmacokinetic parameters of DS-8201a assessed in an earlier Phase 1 trial, 5.4 mg/kg DS-8201a was chosen to assess drug interactions.
Groups:
- Cohort 1: DS-8201a + Ritonavir: Participants who received 5.4 mg/kg DS-8201a as an intravenous infusion once every 3 weeks and 200 mg ritonavir twice daily (BID) on Day 17 of Cycle 2 until Day 21 of Cycle 3.
- Cohort 2: DS-8201a + Itraconazole: Participants who received 5.4 mg/kg DS-8201a as an intravenous infusion once every 3 weeks and 200 mg itraconazole twice daily (BID) on Day 17 of Cycle 2 followed by 200 mg daily (QD) until Day 21 of Cycle 3.
Period: Overall Study
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole
Started | 17 | 23
Completed (Ongoing on study drug as of 26 Sep 2018) | 11 | 19
Not Completed | 6 | 4
Not completed — Progressive disease as per RECIST | 3 | 3
Not completed — Clinical progression | 0 | 1
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: Demographics were assessed in the Safety Analysis Set.
Groups:
- Cohort 1: DS-8201a + Ritonavir: Participants who received 5.4 mg/kg DS-8201a as an intravenous infusion once every 3 weeks and 200 mg ritonavir twice daily on Day 17 of Cycle 2 until Day 21 of Cycle 3.
- Cohort 2: DS-8201a + Itraconazole: Participants who received 5.4 mg/kg DS-8201a as an intravenous infusion once every 3 weeks and 200 mg itraconazole BID on Day 17 of Cycle 2 followed by 200 mg QD until Day 21 of Cycle 3.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.45) | 53.5 (12.91) | 56.5 (11.96)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 10 | 18 | 28
  ≥65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 5 | 13 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 23 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) Following Treatment With DS-8201a and Ritonavir - Cohort 1
Description: Maximum concentration (Cmax) was assessed for DS-8201a and total Anti-HER2 antibody.
Time Frame: Cycle 1: Day 1, pre-dose and end of infusion (EOI); Cycles 2 and 3: Day 1, pre-dose, EOI, 2 hours, 4 hours, 7 hours; Day 2, 4, 8, 12, 17, and 22; Cycles 4, 6 and 8: Day 1, pre-dose and EOI (each cycle is 22 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: DS-8201a + Ritonavir
Number analyzed (Participants) | 12
ug/mL
  DS-8201a, Cycle 2: DS-8201a only | 133 (25.5)
  DS-8201a, Cycle 3: DS-8201a + ritonavir | 140 (23.0)
  Total Anti-HER2 antibody, Cycle 2: DS-8201a only | 121 (22.2)
  Total Anti-HER2 antibody, Cycle 3: DS-8201a + ritonavir | 126 (23.1)

2. Primary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) For MAAA-1181a Following Treatment With DS-8201a and Ritonavir - Cohort 1
Description: Maximum concentration (Cmax) was assessed for MAAA-1181a.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: DS-8201a + Ritonavir
Number analyzed (Participants) | 12
ng/mL
  MAAA-1181a, Cycle 2: DS-8201a only | 8.98 (2.83)
  MAAA-1181a, Cycle 3: DS-8201a + ritonavir | 8.95 (3.68)

3. Primary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve Following Treatment With DS-8201a and Ritonavir - Cohort 1
Description: Area under the serum concentration-time curve from time zero to 17 days (AUC17d) and during the dosing interval (AUCtau) for DS-8201a and total anti-HER2 antibody were assessed.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | Cohort 1: DS-8201a + Ritonavir
Number analyzed (Participants) | 12
ug*d/mL
  DS-8201a, Cycle 2 (DS-8201a only): AUC17d | 650 (168.0)
  DS-8201a, Cycle 2 (DS-8201a only): AUCtau | 701 (185)
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUC17d: number analyzed (Participants) | 8
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUC17d | 754 (137.0)
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUCtau: number analyzed (Participants) | 7
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUCtau | 810 (153.0)
  Total Anti-HER2 antibody, Cycle 2 (DS-8201a only): AUC17d | 723 (191)
  Total Anti-HER2 antibody, Cycle 2 (DS-8201a only): AUCtau | 791 (217)
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUC17d: number analyzed (Participants) | 8
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUC17d | 796 (155)
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUCtau: number analyzed (Participants) | 7
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUCtau | 860 (170)

4. Primary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve of MAAA-1181a Following Treatment With DS-8201a and Ritonavir - Cohort 1
Description: Area under the serum concentration-time curve from time zero to 17 days (AUC17d) and during the dosing interval (AUCtau) were assessed for MAAA-1181a.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | Cohort 1: DS-8201a + Ritonavir
Number analyzed (Participants) | 12
ng*d/mL
  MAAA-1181a, Cycle 2 (DS-8201a only): AUC17d | 32.7 (7.45)
  MAAA-1181a, Cycle 2 (DS-8201a only): AUCtau | 35.0 (8.10)
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUC17d: number analyzed (Participants) | 8
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUC17d | 37.2 (6.93)
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUCtau: number analyzed (Participants) | 7
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUCtau | 39.2 (7.98)

5. Primary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) Following Treatment With DS-8201a and Itraconazole - Cohort 2
Description: Maximum concentration (Cmax) was assessed for DS-8201a and total Anti-HER2 antibody.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Cohort 1: DS-8201a + Itraconazole: Participants who received 5.4 mg/kg DS-8201a as an intravenous infusion once every 3 weeks and 200 mg itraconazole twice daily (BID) on Day 17 of Cycle 2 followed by 200 mg daily (QD) until Day 21 of Cycle 3.
Arm/Group | Cohort 1: DS-8201a + Itraconazole
Number analyzed (Participants) | 14
ug/mL
  DS-8201a, Cycle 2: DS-8201a only | 139 (23.6)
  DS-8201a, Cycle 3: DS-8201a + ritonavir | 142 (23.9)
  Total Anti-HER2 antibody, Cycle 2: DS-8201a only | 119 (19.1)
  Total Anti-HER2 antibody, Cycle 3: DS-8201a + ritonavir | 130 (18.2)

6. Primary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) of MAAA-1181a Following Treatment With DS-8201a and Itraconazole - Cohort 2
Description: Maximum concentration (Cmax) was assessed for MAAA-1181a.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 14
ng/mL
  MAAA-1181a, Cycle 2: DS-8201a only | 8.65 (2.03)
  MAAA-1181a, Cycle 3: DS-8201a + ritonavir | 8.93 (1.77)

7. Primary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve Following Treatment With DS-8201a and Itraconazole - Cohort 2
Description: Area under the serum concentration-time curve from time zero to 17 days (AUC17d) and during the dosing interval (AUCtau) were assessed for DS-8201a and total anti-HER2 antibody.
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 14
ug*d/mL
  DS-8201a, Cycle 2 (DS-8201a only): AUC17d | 644 (188)
  DS-8201a, Cycle 2 (DS-8201a only): AUCtau | 706 (211)
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUC17d | 710 (187)
  DS-8201a, Cycle 3 (DS-8201a + ritonavir): AUCtau | 789 (217)
  Total Anti-HER2 antibody, Cycle 2 (DS-8201a only): AUC17d | 707 (194)
  Total Anti-HER2 antibody, Cycle 2 (DS-8201a only): AUCtau | 790 (224)
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUC17d | 781 (196)
  Total Anti-HER2 antibody, Cycle 3 (DS-8201a + ritonavir): AUCtau | 883 (238)

8. Primary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve of MAAA-1181a Following Treatment With DS-8201a and Itraconazole - Cohort 2
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 14
ng*d/mL
  MAAA-1181a, Cycle 2 (DS-8201a only): AUC17d | 29.9 (8.31)
  MAAA-1181a, Cycle 2 (DS-8201a only): AUCtau | 32.4 (9.21)
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUC17d | 34.8 (8.04)
  MAAA-1181a, Cycle 3 (DS-8201a + ritonavir): AUCtau | 37.7 (8.87)

9. Secondary Outcome: Best Objective Response as Confirmed By The Investigator's Assessment in Participants With HER2-Expressing Advanced Solid Malignant Tumors
Description: Best objective response (BOR) was assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Completed response (CR) was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline up to disease progression, death, lost to follow up, or study discontinuation (whichever comes first), up to approximately 9 months post-dose
Population: Response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 17 | 19
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 9 | 10
  Stable disease (SD) | 8 | 8
  Non-CR/Non-PR | 0 | 0
  Progressive disease (PD) | 0 | 1
  Non evaluable | 0 | 0

10. Secondary Outcome: Objective Response Ratio (ORR) as Confirmed By The Investigator's Assessment in Participants With HER2-Expressing Advanced Solid Malignant Tumors
Description: Objective response ratio (ORR) was defined as the proportion of participants who achieved CR and PR as assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 9
Population: Response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 17 | 19
Participants | 9 | 10

11. Secondary Outcome: Objective Response Rate as Confirmed By The Investigator's Assessment in Participants With HER2-Expressing Advanced Solid Malignant Tumors
Description: Objective response rate (defined as participants who achieved CR and PR) was assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. ORR with confirmation is Objective Response Rate applying a confirmed response of CR/PR in RECIST version 1.1.
Time Frame: as for outcome 9
Population: Response was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole
Number analyzed (Participants) | 17 | 19
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to approximately 9 months post-dose.
Arm/Group | Cohort 1: DS-8201a + Ritonavir | Cohort 2: DS-8201a + Itraconazole
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/17 | 3/23
Other Adverse Events (participants affected / at risk) | 17/17 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-8201a + Ritonavir (N=17) | Cohort 2: DS-8201a + Itraconazole (N=23)
Disease progression (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-8201a + Ritonavir (N=17) | Cohort 2: DS-8201a + Itraconazole (N=23)
Nasopharyngitis (Infections and infestations) | 3 | 0
Paroncyhia (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 2
Dysgeusia (Nervous system disorders) | 1 | 1
Akathisia (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 15
Constipation (Gastrointestinal disorders) | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 3 | 8
Stomatitis (Gastrointestinal disorders) | 4 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Fatigue (General disorders) | 5 | 4
Malaise (General disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 8
White blood cell count decreased (Investigations) | 7 | 7
Platelet count decreased (Investigations) | 9 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 5
Alanine aminotransferase increased (Investigations) | 7 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Weight decreased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 2 | 1
Troponin I increased (Investigations) | 1 | 1
Alanine aminotransferase decreased (Investigations) | 1 | 0
Aspartate aminotransferase decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Ophthalmological examination abnormal (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT03383692/Prot_SAP_000.pdf